CLINICAL TRIAL: NCT00568646
Title: A Phase 2 Study of Oral MKC 1, Administered Twice Daily for 14 Consecutive Days in a 28-Day Cycle, in Patients With Unresectable or Metastatic Pancreatic Cancer Who Have Failed at Least One Prior Chemotherapy Regimen in Either the Neoadjuvant, Adjuvant, or First-line Metastatic Setting
Brief Title: Phase 2 Study of Oral MKC-1 in Patients With Unresectable or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Carolyn Sidor, Miikana Therapeutics, an EntreMed, Inc. Company
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-105
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MKC-1

INTERVENTIONS:
Drug: MKC-1 — Oral MKC-1 capsules, administered twice daily, for 14 consecutive days, in a 28-day cycles

SUMMARY:
To determine the antitumor activity of MKC-1 in patients with unresectable or metastatic pancreatic cancer who have failed at least one prior chemotherapy regimen in either the neoadjuvant, adjuvant, or first-line metastatic setting

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and Health Insurance Portability and Accountability Act authorization for release of protected health information before any study related assessments
* Have histologically confirmed pancreatic cancer and measurable disease according to RECIST
* Have failed at least one prior chemotherapy regimen in either the neoadjuvant, adjuvant, or first-line metastatic setting
* Be at least 18 years of age at the time of consent
* Have an Eastern Cooperative Oncology Group performance status of 0 or 1
* Have the following laboratory results, within 10 days before the first MKC 1 administration:

  1. Hemoglobin greater than or equal to 9 g/dL
  2. Absolute neutrophil count greater than or equal to 1.5 x 109 cells/L
  3. Platelet count greater than or equal to 75 x 109 cells/L
  4. Serum creatinine less than or equal to 1.5 times the upper limit of normal (ULN)
  5. Aspartate transaminase less than or equal to 2.5 times the ULN
  6. Serum albumin greater than or equal to 3.0 g/dL
  7. Total bilirubin less than or equal to the ULN

Exclusion Criteria:

* Be a pregnant or breast-feeding woman. Female patients must be postmenopausal, surgically sterile, or they must agree to use a barrier method of contraception. Female patients of childbearing potential must have a negative pregnancy test within the 10 days before the first MKC 1 administration. Male patients must be surgically sterile or agree to use an acceptable method of contraception.
* Have known central nervous system metastases unless they are being treated, are clinically stable, and do not require the use of steroids.
* Have clinical evidence of significant bowel obstruction, active uncontrolled malabsorption syndromes, or a history of total gastrectomy.
* Have uncontrolled hypercalcemia (serum calcium-corrected greater than 12 mg/dL).
* Have a serious cardiac condition (Class III/IV congestive heart failure according to New York Heart Association classification) or documented acute myocardial infarction within the previous 6 months.
* Have any medical conditions that, in the investigator's opinion, would impose excessive risk to the patient. These conditions include: infection requiring parenteral or oral anti-infective treatment or any altered mental status or any psychiatric condition that would interfere with the understanding of the informed consent.
* Have had previous malignancies, unless free of recurrence for at least 5 years except cured basal cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix.
* Be receiving treatment with antiretroviral therapy metabolized through CYP3A4 (including indinavir, nelfinavir, ritonavir, and saquinavir, or any other medications that interfere with CYP3A4).
* Have, in the opinion of the investigator, any clinically significant existing toxicities from previous chemotherapy therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate based on tumor measurements according to the RECIST | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Kwak, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Faris JE, Arnott J, Zheng H, Ryan DP, Abrams TA, Blaszkowsky LS, Clark JW, Enzinger PC, Hezel AF, Ng K, Wolpin BM, Kwak EL. A phase 2 study of oral MKC-1, an inhibitor of importin-beta, tubulin, and the mTOR pathway in patients with unresectable or metastatic pancreatic cancer. Invest New Drugs. 2012 Aug;30(4):1614-20. doi: 10.1007/s10637-011-9708-3. Epub 2011 Jul 29. PMID 21800081